CLINICAL TRIAL: NCT07259733
Title: Strategy for Rapid Control of Apparent Resistant Arterial Hypertension in the Public Health System (FAST Control)
Brief Title: Rapid Management of Resistant Hypertension in the Public Health System (Fast Control)
Acronym: FastControl
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Collaborators: Servier (Industry)
Responsible Party: Principal Investigator, Fabrizio Urbinati Maroja, MD, MSc, Instituto Dante Pazzanese de Cardiologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 56042422900005462
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Apparent Resistant Hypertension; Hypertension; High Blood Pressure
Keywords: Apparent resistant hypertension; Fixed-dose combination; Triple combination therapy; Perindoprile; Indapamide; Amlodipine; Clinical Trial; Brazil
MeSH Terms: conditions — Hypertension | interventions — Indapamide; Amlodipine

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 1:1 ratio to receive either a simplified fixed-dose triple combination (perindopril 10 mg/indapamide 2.5 mg/amlodipine 10 mg once daily) or usual care with their current individualized antihypertensive regimen (up to five drug classes). Each group follows its assigned treatment throughout the 12-week study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simplified Fixed-Dose Triple Combination (Experimental): Randomized participants in this group discontinue their previous antihypertensive medications and replace them with the single-pill triple fixed-dose combination. Treatment adjustments may be made if required according to office blood pressure measurements.
  Interventions: Drug: Triple Fixed-Dose Combination (Perindoprile/Indapamide/Amlodipine)
- Usual Care Antihypertensive Regimen (Active Comparator): Participants continue their usual antihypertensive treatment regimen, consisting of up to five drug classes administered as separate tablets, for 12 weeks, with medication adjustments performed as needed according to office blood pressure measurements.
  Interventions: Drug: Usual Care Antihypertensive Regimen

INTERVENTIONS:
Drug: Triple Fixed-Dose Combination (Perindoprile/Indapamide/Amlodipine) — Participants receive a fixed-dose tablet containing perindopril 10 mg, indapamide 2.5 mg, and amlodipine 10 mg administered once daily for 12 weeks. Randomized participants in this group discontinue their previous antihypertensive medications and replace them with the single-pill triple fixed-dose combination. Treatment adjustments may be made if required according to office blood pressure measurements
  Arms: Simplified Fixed-Dose Triple Combination
Drug: Usual Care Antihypertensive Regimen — Participants continue their usual antihypertensive therapy, consisting of up to five drug classes administered as separate tablets. Medication types and doses are adjusted by the investigator as needed to achieve office blood pressure control, following standard clinical practice. Treatment modifications are permitted throughout the 12-week study period according to clinical judgment and blood pressure response.
  Arms: Usual Care Antihypertensive Regimen

SUMMARY:
This is a single-center, open-label, randomized clinical trial conducted at the Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil. The study evaluates a simplified treatment strategy for patients with apparent resistant hypertension, comparing fixed triple combination therapy (perindopril, indapamide, and amlodipine) with usual care using multiple separate antihypertensive drugs. The primary objective is to compare 24-hour blood pressure control as measured by ABPM at 12 weeks between the two treatment strategies. Enrollment began on July 15, 2023, and this study was registered retrospectively.

DETAILED DESCRIPTION:
Resistant hypertension remains a major clinical challenge, frequently resulting from therapeutic inertia, poor adherence, and the complexity of multi-drug regimens. Simplified treatment strategies, such as fixed-dose combinations, have been proposed to improve adherence and blood pressure control.

The FAST Control study is a single-center, open-label, randomized (1:1), parallel-group clinical trial designed to compare the efficacy of a simplified treatment strategy versus usual care in patients with apparent resistant hypertension (aRHTN). The simplified treatment consists of a fixed triple combination of perindopril 10 mg, indapamide 2.5 mg, and amlodipine 10 mg once daily, while the usual care group maintains their current regimen with up to five antihypertensive drug classes administered as separate tablets.

Eligible participants are adults aged 18 to 75 years, followed at the Hypertension Section of the Instituto Dante Pazzanese de Cardiologia (São Paulo, Brazil), presenting with uncontrolled blood pressure despite treatment with 3-5 drug classes (including a renin-angiotensin system blocker, a thiazide or thiazide-like diuretic, and a long-acting calcium channel blocker). Apparent resistant hypertension is confirmed by 24-hour ambulatory blood pressure monitoring (ABPM) showing a mean BP ≥130/80 mmHg. Participants with secondary hypertension, severe comorbidities, or contraindications to the study medications are excluded.

The primary objective is to compare the rate of 24-hour blood pressure control as measured by ABPM at 12 weeks between the simplified treatment and usual care groups. Secondary objectives include evaluating the difference in absolute reduction of 24-hour blood pressure (BP), as measured by ABP between the two groups; comparing the office blood pressure control rate after 12 weeks between the groups; assessing the difference in absolute reduction of office blood pressure between the groups; and comparing the number of antihypertensive drug classes and the total number of pills used between the groups throughout the study.

This study was approved by the Research Ethics Committee of the Instituto Dante Pazzanese de Cardiologia (CAAE [56042422900005462]) and registered retrospectively, as patient enrollment began on July 15, 2023.

ELIGIBILITY:
Inclusion Criteria: Age between 18 and 75 years;

Treatment with 3 to 5 classes of antihypertensive drugs, including a maximum dose of an ACE inhibitor or ARB, a thiazide or thiazide-like diuretic, and a calcium channel blocker (CCB);

Recent 24-hour ambulatory blood pressure monitoring (ABPM) (<1 month) showing values above target (24-hour BP ≥130/80 mmHg);

Office blood pressure ≥140/90 mmHg;

Poor adherence to treatment, defined as a score ≥1 point on the Morisky Medication Adherence Scale (MMAS-4).

-

Exclusion Criteria:Secondary hypertension (including hyperaldosteronism, pheochromocytoma, or renovascular hypertension);

History of intolerance or adverse reactions to study medications, such as ACE inhibitors (cough or angioedema), thiazide or thiazide-like diuretics (electrolyte disturbances), or calcium channel blockers (significant ankle edema or headache);

Indispensable use of beta-blockers or mineralocorticoid receptor antagonists;

Office blood pressure ≥ 220 × 120 mmHg;

Reduced left ventricular ejection fraction (LVEF < 55%);

Severe renal impairment (creatinine clearance < 30 mL/min or eGFR < 30 mL/min/1.73 m²);

Atrial fibrillation or atrial flutter;

Use of oral anticoagulants;

Significant valvular heart disease;

Body mass index (BMI) ≥ 40 kg/m²;

Pregnant or breastfeeding women;

Severe psychiatric disorders;

Active malignancy with life expectancy < 2 years;

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of 24-hour Blood Pressure Control Measured by ABPM at 12 weeks | 12 weeks
  Proportion of participants achieving 24-hour mean blood pressure <130/80 mmHg, as measured by ambulatory blood pressure monitoring (ABPM), after 12 weeks of treatment.
Rate of 24-hour Blood Pressure Control Measured by Ambulatory Blood Pressure Monitoring (ABPM) at 12 weeks | 12 weeks
  Proportion of participants achieving 24-hour mean blood pressure <130/80 mmHg, as measured by ambulatory blood pressure monitoring (ABPM), after 12 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the primary and secondary outcome measures will be shared after de-identification. Data will be available upon reasonable request to qualified researchers for purposes of verification or secondary analysis.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: December, 2026
Access Criteria: Participants data and supporting documents will be available to qualified researchers for scientific purposes upon reasonable request. Access will be granted after approval of a written proposal and execution of a data use agreement. Data will be shared eletronically through secure institutional channels.